CLINICAL TRIAL: NCT06056596
Title: Intra-ocular Penetration of Oral Lamivudine and Measurement of Systemic Inflammatory Markers in Patients Undergoing Rhegmatogenous Retinal Detachment Surgery
Brief Title: Lamivudine and Plasma Markers of Inflammation in Retinal Detachment
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Treatment approach changed, and insufficient population
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-1223; SMPH/OPHTHAL&VIS SCI/FPRC (Other: UW Madison); Protocol Version 1/29/2024 (Other: UW Madison)
Record Dates: First submitted 2023-08-01; First posted 2023-09-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Retinal Detachment; Rhegmatogenous Retinal Detachment
Keywords: vitrectomy surgery
MeSH Terms: conditions — Retinal Detachment | interventions — Lamivudine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lamivudine (Experimental): Lamivudine 300mg PO once daily for three days
  Interventions: Drug: Lamivudine 300 MG
- Placebo (Placebo Comparator): Placebo once daily for three days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lamivudine 300 MG — Drug to be taken once daily for three days (two days prior to surgery and on the morning of surgery)
  Arms: Lamivudine
Drug: Placebo — Dose to be taken once daily for three days (two days prior to surgery and on the morning of surgery)
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to test whether an oral medication (lamivudine) enters the eye and reduces blood markers of inflammation in people who undergo retinal detachment surgery (pars plana vitrectomy).

Participants will take the study medication or placebo, and the researchers will measure blood markers of inflammation before and after surgery. The researchers will also measure the amount of medication in the blood and fluid inside the participant's eye (which is collected during surgery).

DETAILED DESCRIPTION:
Lamivudine is an anti-viral medication that has intrinsic anti-inflammatory properties that could be useful in the treatment of vitreoretinal disease. It is not known whether lamivudine enters the eye after oral administration. The purpose of this study is to measure the intra-ocular concentration of lamivudine after oral administration in participants that require pars plana vitrectomy surgery for repair of rhegmatogenous retinal detachment. Participants undergoing retinal detachment surgery will receive oral lamivudine for three days prior to surgery; lamivudine will be measured intra-operatively (vitreous and aqueous humor) and pre-operatively (plasma). Plasma markers of inflammation will be measured before and after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 or ≤ 75 years
* Patients with rhegmatogenous retinal detachment that require vitrectomy surgery

Exclusion Criteria:

* Previous pars plana vitrectomy in the affected eye
* Positive for Hepatitis B surface antigen or HIV antibodies, or history of Hepatitis B/HIV
* Pregnant or breast-feeding
* Liver disease or abnormal AST/ALT
* Renal impairment (Creatinine clearance < 50)
* Diabetes with current use of insulin
* Anemia (Hemoglobin <13.2 g/dL (male) or < 11.6 g/dL (female))
* Unwilling to hold concurrent use of sorbitol or sorbitol-containing medications or products while taking study medication(including, but not limited to: blackberries, raspberries, strawberries, stone fruits, apples, avocados, sugar-free items such as chewing gum, hard candies, snack bars, frozen desserts, and chocolates, liquid and capsule/caplet analgesics, cough/cold/flu syrup, liquid and capsule/caplet pseudoephedrine, chewable antacid tablets, liquid and capsule allergy medications, motion sickness and nausea medications)
* Current use of trimethoprim-sulfamethoxazole
* Pancreatitis or history of pancreatitis
* Uncontrolled blood pressure (> 160 mm Hg systolic or >100 mm Hg diastolic) within the last 3 months, or current use of more than one anti-hypertensive medication
* History of stroke, myocardial infarction, or congestive heart failure
* Current vitreous hemorrhage that obscures view of retinal details
* Patients with a shallow anterior chamber or in whom anterior chamber paracentesis is considered unsafe

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-06 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of lamivudine after oral administration | Pre-operative
  Mean concentration of lamivudine in plasma
Intra-ocular concentration of lamivudine after oral administration | Intra-operatively
  Mean concentration of lamivudine in vitreous and aqueous humor

SECONDARY OUTCOMES:
Change in erythrocyte sedimentation rate (millimeter per hour) | Pre-operative to one week post-operative
  Mean concentration of inflammatory markers will in part be measured by erythrocyte sedimentation rate.
Change in C-reactive protein (milligrams per liter) | Pre-operative to one week post-operative
  Mean concentration of inflammatory markers will in part be measured by C-reactive protein.
Change in concentration of inflammatory markers (picogram per milliliter) | Pre-operative to one week post-operative
  Mean concentration of inflammatory markers will in part be measured by tumor necrosis factor alpha, interleukin (IL)-18, IL-1 beta, IL-6, IL-10, MCP-1, MIP-1 alpha, GM-CSF in picograms per milliliter.
Change in concentration of inflammatory markers (micrograms per milliliter) | Pre-operative to one week post-operative
  Mean concentration of inflammatory markers will in part be measured by interferon (IFN) alpha, IFN beta, IFN gamma in micrograms per milliliter)
Change in concentration of soluble IL-2 receptor alpha (Units per milliliter) | Pre-operative to one week post-operative
  Mean concentration of inflammatory markers will in part be measured by soluble IL-2 receptor alpha in Units per milliliter.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Altaweel, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes